CLINICAL TRIAL: NCT03524820
Title: Cetuximab Monotherapy or Cetuximab + Chemotherapy for Third Line Rechallenge in Metastatic Colorectal Cancer, RAS+ (RAt Sarcoma Gene) Wild Type Patients, Who Were Treated With Cetuximab Chemotherapy as First Line Treatment
Brief Title: Cetuximab Therapy for Third Line Rechallenge in Metastatic Colorectal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: By Merck
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Merck Serono International SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0436-17
Record Dates: First submitted 2018-03-07; First posted 2018-05-15 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2021-02

CONDITIONS: Cancer of Colon
Keywords: cetuximab, colon cancer, RAS
MeSH Terms: conditions — Colonic Neoplasms | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Metastatic colorectal cancer patients (Experimental): Metastatic colorectal cancer patients receiving third line cetuximab treatment
  Interventions: Drug: Cetuximab

INTERVENTIONS:
Drug: Cetuximab — Administration of drug
  Other Names: Erbitux

SUMMARY:
This research is intended to check the benefit of treatment with cetuximab in metastatic colorectal cancer patients with wild type RAS as third line treatment. The advantage to the patients is unclear. This study will look if mutations in patients' blood area predictive marker for progression free time (FPT) in metastatic colorectal cancer patients treated with third line cetuximab. A predictive marker for FPT metastatic colorectal cancer patients treated with third line cetuximab will enable a reduction in the number of treated patients. Treatment only of patients with a positive marker is expected to prevent inefficient treatment which will reduce suffering for the patients and reduce unnecessary medical treatment.

DETAILED DESCRIPTION:
This research is intended to check the benefit of treatment with cetuximab in metastatic colorectal cancer patients with wild type RAS as third line treatment, following first line cetuximab treatment and other second line treatments. The hypothesis is that most cetuximab sensitive cells will be eliminated in the first line of treatment, but may reemerge following other second line treatments which are targeted to other clones in the tumor. The advantage to the patients is unclear, however some preliminary studies show advantage to patients. This study will look if mutations in patients' blood are a predictive marker for progression free time (FPT) in metastatic colorectal cancer patients treated with third line cetuximab. A predictive marker for FPT metastatic colorectal cancer patients treated with third line cetuximab will enable a reduction in the number of treated patients. Treatment only of patients with a positive marker is expected to prevent inefficient treatment which will reduce suffering for the patients and reduce unnecessary medical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 18
* Tissue diagnosis of metastatic colon cancer without operational or radiation therapy options
* No RAS mutation in tumor tissue
* Measurable disease according to RACIST criteria v1.1
* ECOG ( Eastern Cooperative Oncology Group) performance status <=2
* Life expectancy of over 3 months
* Women of fertility age not pregnant
* Ability to understand and sign and informed consent form to participate in the trial and the ability to perform the treatment and follow up required for participation in the trial
* At least three months progression free time in first line cetuximab treatment
* Disease progression according to RACIST v1.1 for first and second lines
* Third line treatment will be applied no less then 17 weeks following and of first line treatment

Exclusion Criteria:

* RAS mutation carriers, or patients with uncertain metastatic colon cancer diagnosis
* Patients operated two weeks prior to accepting trail drug, or that did not recover from treatment
* Level 3 allergic response to any of trial drugs
* First line cetuximab treatment stopped due to allergic response
* Severe medical or mental diagnosis which might increase the risk in drug administration according to treating physician's discretion
* Pregnant or lactating women

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-10-17 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
response to treatment | 5 years
  CT based on standard RECIST criteria

CONTACTS AND LOCATIONS:
Overall Officials: Aviad Zick, MD PhD, Principal Investigator — Senior medical oncologist, Head of Cancer Genetics Laboratory, Dep. of Oncology
Locations (1):
- Hadassah Ein Kerem, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No